CLINICAL TRIAL: NCT06140485
Title: A Phase III, Randomized, Double-Blind, Double-Dummy, Active- Controlled Clinical Trial to Investigate the Efficacy and Safety of NW Low-Glu® in Patients With Type II Diabetes Mellitus
Brief Title: A Trial to Investigate the Efficacy and Safety of NW Low-Glu® in Patients With Type II Diabetes Mellitus
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Natural Wellness Egypt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NW_LowGlu_18052023
Record Dates: First submitted 2023-11-12; First posted 2023-11-20 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes mellitus; Complementary medicine; Alternative medicine
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NW Low-Glu® (Experimental): Patients in this arm will receive one placebo tablet plus two NW Low-Glu® capsules administered PO on empty stomach with plenty of water 2 hours after meals twice daily.
  A total dose of four NW Low-Glu® capsules will be administered per day.
  Interventions: Dietary Supplement: NW Low-Glu®
- Metformin (Active Comparator): Patients in this arm will receive one metformin 1000 mg tablet plus two placebo capsules administered PO on an empty stomach with plenty of water 2 hours after meals twice daily.
  A total dose of Metformin 2000 mg will be administered per day.
  Interventions: Drug: Metformin

INTERVENTIONS:
Dietary Supplement: NW Low-Glu® — One NW Low-Glu® capsule contains Mas Cotek powdered Extract 300 mg (from leaves of Ficus deltoidea Jack by aqueous solvent extraction) + Cinnamomum cassia L. powdered Extract 100 mg + Black seed powdered extract 250 mg (from seeds of Nigella sativa L. by 70% hydro-alcoholic extraction).
  Arms: NW Low-Glu®
Drug: Metformin — Patients in the active comparator arm will receive a total of 2000 mg of metformin per day.
  Arms: Metformin

SUMMARY:
The goal of this clinical trial is to investigate efficacy and safety of an herbal medicinal product of (NW Low-Glu®) in patients with Type 2 Diabetes Mellitus (T2DM). The main question[s] it aims to answer are:

• What will be the mean change in HbA1c levels in the experimental arm (NW Low-Glu®) compared to the active-control arm (metformin) after 6 months of treatment?

Participants will randomized in a 1:1 allocation ratio, into one of the two treatment groups, to receive either Metformin or NW Low-Glu®.

Researchers will compare the mean change in HbA1C, fasting blood glucose, and weight between the experimental arm and the active-control arm.

DETAILED DESCRIPTION:
Despite the advancements in drug discovery and the increase in the total budget spent on pharmaceutical research and development, the number of new drug approvals has decreased in the recent years. Not only do plants serve as foods, but they have also been an integral part of therapeutic interventions in traditional and alternative medicine throughout human history. Because plants comprise a large number of monomeric compounds, herbal medicine continues to play a multi-targeted approach role in treating diseases.

It is estimated that 25% of modern drugs are derived from natural products. In addition, the World Health Organization (WHO) estimates that between 65% and 80% of developing countries use medicinal plants as remedies. In a study conducted in Alexandria, Egypt, the rate of using complementary and alternative medicine (CAM) at least once among type 2 diabetes mellitus (T2DM) patients was 41.7%, with 26.3% being regular CAM users. The main reason for resorting to CAM was the belief in its benefits. The powdered extracts of Ficus deltoidea leaves, Cinnamomum cassia bark, and Nigella Sativa seeds (Black Seeds) have been used for the treatment of diabetes and other medical conditions for over 2000 years. Studies on the individual effect of each of these medicinal plants have demonstrated antihyperglycemic efficacy in individuals with T2DM. For example, Kalman et al. reported significant reduction in glucose and lipid levels upon testing the antidiabetic effects of F. deltoidea in adults with prediabetes. There is also strong evidence to support the efficacy of Cinnamomum cassia in lowering fasting plasma glucose (FPG). In a randomized controlled trial, poorly controlled T2DM patients receiving an aqueous extract equivalent to 3 grams of Cinnamomum cassia for 4 months had significantly higher reduction in FPG compared to placebo (10.3% vs 3.4%). Furthermore, Nigella Sativa seeds' extract (in combination with oral hypoglycemic drugs) led to significant reductions in FPG, 2-hour post-prandial glucose (2 hr PPG), HbA1c, and insulin resistance at 12 weeks, which makes it a possible beneficial adjuvant therapy to oral hypoglycemics in patients with uncontrolled T2DM. A combination of the mentioned medicinal herbs is registered as NW Low-Glu® (a dietary supplement; one capsule constitutes 300 mg Mas Cotek powdered extract [from leaves of Ficus deltoidea Jack by aqueous solvent extraction] + 100 mg Cinnamomum cassia L. powdered extract +250 mg Black Seed powdered extract [from seeds of Nigella sativa L. by 70% hydro-alcoholic extraction]) in the Malaysian market under the registration number MAL15070037 T.

The efficacy and safety NW Low-Glu® was investigated in a phase II study in 2022, in which the hypoglycemic effect of two doses of the herbal medicinal product was compared in patients newly diagnosed with T2DM. Correspondingly, the results of the phase II study warranted further assessment of NW Low-Glu® activity in patients inclined to benefit from it.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following criteria to be eligible for enrolment into the study.

1. Able and willing to provide written informed consent.
2. Male and female patients aged between 18 and 65 years.
3. Recently diagnosed patients with T2DM (within two years prior to enrollment).
4. Patients with dysglycemia with HbA1c of 5.7%-8.7%.
5. Treatment-naïve patients OR patients who discontinued their anti-diabetic medications within three months prior to enrollment.

Exclusion Criteria:

Patients meeting any of the following criteria are not eligible for enrolment into the study.

1. Pregnant or lactating women; women of childbearing potential must agree to use an accepted method of contraception during the course of the study and for one month after their last dose of study drug.
2. Patients with BMI > 40 Kg/m2 or BMI < 18.5 Kg/m2.
3. Estimated glomerular filtration rate (eGFR) <60 mL/min/1.73 m2 (measured by the Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] equation).
4. History of positive human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAG), or hepatitis C (HCV) antibody test.
5. History of type I diabetes, diabetes resulting from pancreatic injury, or secondary forms of diabetes such as Cushing's syndrome or acromegaly.
6. History of diabetic complications such as diabetic ketoacidosis, lactic acidosis or state of hyperosmolar hyperglycemia, diabetic proliferative retinopathy, or severe diabetic neuropathy (requiring treatment with antidepressants or opioids) and history of decompensated diabetes (polyuria, polydipsia, nocturia, fatigue).
7. History of chronic gastrointestinal (GI) conditions that could impede gastric emptying or potentially affect the interpretation of the study data.
8. History of weight loss surgery or weight loss procedure involving the GI tract, such as gastric bypass, gastric stapling, or gastric banding.
9. History of an eating disorder (e.g., bulimia, anorexia).
10. History of malignancy (except treated basal or squamous cell skin cancer) within five years prior to screening.
11. History of significant cardiovascular disease (such as congestive heart failure, myocardial infarction, coronary disease) or uncontrolled hypertension.
12. History of clinically significant renal or liver disease.
13. Receipt of an investigational drug within 30 days prior to screening, or active enrollment in another investigational medication or device trial.
14. Known or suspected allergy to the trial products.
15. Any condition, in the judgment of the investigator, that would interfere with the patient's ability to comply with all study requirements or that would place the patient at unacceptable risk by his/her participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Comparing the mean change in HbA1c levels between the experimental arm and the active-control arm | 6 months
  To compare the hypoglycemic effect of a herbal medicinal product (NW Low-Glu) to that of metformin as measured by the mean change in HbA1c levels in patients with type II diabetes mellitus.

SECONDARY OUTCOMES:
Comparing the mean change in HbA1c levels between the experimental arm and the active-control arm Comparing the mean change in fasting blood glucose levels | 6 months
  To compare the hypoglycemic effect of a herbal medicinal product (NW Low-Glu) to that of metformin as measured by the mean change in fasting blood glucose levels in patients with type II diabetes mellitus.
Measuring the incidence of AEs, SAEs, TEAEs, hypoglycemic events, and abnormal laboratory test findings in both the experimental arm and the active comparator arm | 6 months
  To measure the incidence of adverse events (AEs), serious adverse events (SAEs), treatment-emergent adverse events (TEAEs), hypoglycemic events, and abnormal laboratory test findings in both the experimental arm and active comparator arm
Assessing cardiovascular AEs in both the experimental arm and the active comparator arm | 6 months
  To measure the number, nature, and severity of cardiovascular AEs and their causal relationship to the received intervention in both the experimental arm and active comparator arm
Comparing the mean change in weight between the experimental arm and the active-control arm | 6 months
  To compare the mean change in body weight between the experimental arm and the active comparator arm

IPD SHARING:
Plan to Share IPD: No